CLINICAL TRIAL: NCT06711198
Title: The Effect of Virtual Reality Simulation on Self-Efficacy and Anxiety Levels of Students in Episiotomy Education: a Randomized Controlled Trial
Brief Title: Virtual Reality Simulation in Episiotomy Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, yasemin hamlacı başkaya, Assoc. prof., Sakarya University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 16112024
Record Dates: First submitted 2024-11-26; First posted 2024-12-02 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Episiotomy; Virtual Simulation
Keywords: virtual simulation; midwifery; episiotomy; anxiety; Self-Efficacy
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: The control group, the calf tongue group, will have an episiotomy on the calf tongue. The virtual reality group will have an episiotomy with virtual reality glasses. The mixed group will first have an episiotomy on the calf tongue with virtual reality glasses and then have an episiotomy on the calf tongue.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control group (application with calf tongue) (No Intervention): Control group (application with calf tongue): In Sakarya University Midwifery Department, while teaching episiotomy application within the scope of Normal birth and postpartum period course, laboratory application is routinely performed on calf tongue. Therefore, the application group to be performed on calf tongue was accepted as the control group. The instructor will first provide theoretical training on episiotomy to the group coming to the laboratory. The theoretical training period will consist of 50 minutes. The content of the training will include the importance of episiotomy, risks, indications, contraindications, episiotomy application time, materials used, episiotomy types, episiotomy repair and time, suture techniques and midwifery care in episiotomy. While explaining suture techniques within the scope of this course, videos about suture techniques on social media platforms will be watched by students. Immediately after the training, episiotomy repair (suture techniques) ap
- 1. Experimental group (Application with virtual reality simulation) (Experimental): The instructor will first provide theoretical training to the group coming to the laboratory on episiotomy. The theoretical training will consist of 50 minutes. The content of the training will include the importance of episiotomy, risks, indications, contraindications, episiotomy application time, materials used, episiotomy types, episiotomy repair and time, suture techniques and midwifery care in episiotomy. While explaining suture techniques within the scope of this course, videos on suture techniques on social media platforms will be watched by the students. Immediately after the training, the episiotomy repair (suture techniques) application will be started. Students will be taken to the laboratory one by one. The student who is taken to the application will be put on the Meta Quest 3 virtual reality glasses and the episiotomy application will be started via the computer integrated with the glasses. The episiotomy application will start with the image of a woman who has given bir
  Interventions: Other: virtual reality simulation
- 2. Experimental group (Both calf tongue and virtual reality simulation) (Experimental): Students in this group will first receive theoretical training as in other groups. The theoretical training will consist of 50 minutes. The content of the training will include the importance of episiotomy, risks, indications, contraindications, episiotomy application time, materials used, episiotomy types, episiotomy repair and time, suture techniques and midwifery care in episiotomy. While suture techniques are explained in this course, videos about suture techniques on social media platforms will be watched by students. Immediately after the training, an application will be made in a virtual reality simulation for episiotomy repair, and then the application will be repeated on the calf tongue.
  Interventions: Other: virtual reality simulation

INTERVENTIONS:
Other: virtual reality simulation — The student will be put on the Meta Quest 3 virtual reality glasses and the episiotomy application will be started via the computer integrated with the glasses. The episiotomy application will start with the image of a woman who has given birth in the delivery room on the delivery table. The student is expected to select the appropriate materials and complete the episiotomy repair of the woman with the correct steps.
  Arms: 1. Experimental group (Application with virtual reality simulation); 2. Experimental group (Both calf tongue and virtual reality simulation)

SUMMARY:
The correct application and repair of episiotomy, which is a frequently used intervention in labor, is important for the psychological and physiological health of the mother after birth. Therefore, it is very important to provide students with the skill of performing episiotomy with the most effective education methods, to reduce their anxiety in this regard and to increase their self-efficacy. Trying to teach suture techniques on sponge, chicken, calf tongue or a soft material is quite limited when the integrity of episiotomy education is considered. Developments in simulation techniques, especially virtual reality glasses that help users experience sensory information such as visual, auditory and movement with real-like experiences, reveal the importance of using technology in health education. Since it does not require additional materials such as calf tongue, sponge, needle holder, etc., it is important for midwifery education to be economical. In addition, the fact that the application can be repeated many times without harming the person affects the anxiety and self-efficacy levels of students before real clinical experience. Within the scope of the study, in order to evaluate the effect of using virtual reality in teaching episiotomy application and repair on students' episiotomy self-efficacy and anxiety levels, midwifery students taking the Normal Birth and Postpartum period course will be divided into three groups during the episiotomy teaching application; one group will practice on calf tongue, one group will practice only with virtual reality, and one group will practice using both. The study data will be collected through the Student Identification Form, State Anxiety Inventory, and Episiotomy Self-Efficacy Scale. The analysis of the data obtained from the research will be done with the SPSS program. It is thought that the study will make a significant contribution to the literature in terms of evaluating the effect of virtual reality glasses on episiotomy teaching.

DETAILED DESCRIPTION:
Episiotomy, which is among the duties of midwives, is an important surgical incision made in the vagina and perineum to widen the vaginal opening during birth (Hersh & Emeis, 2020). In many countries, especially those classified as low or middle income; the majority of women who give birth vaginally undergo routine episiotomy (Silf et al. 2015). Although the use of routine episiotomy is no longer recommended, a midwife or obstetrician must perform the procedure expertly (Güler et al. 2018). Correct application and repair of episiotomy is important for the psychological and physiological health of the mother after birth. If this process is not managed correctly, it can reduce the quality of life of women (Güler et al. 2018, Demir Kaymak et al., 2024). For this reason, it is very important to provide students with the skill of performing episiotomy with the most effective training methods and to increase their self-efficacy in this regard (Bick et al., 2010; Güler et al. 2018). Virtual reality is a simulation technology that allows people to feel like they are in a real world through technological tools using three-dimensional images made in a computer environment, and allows them to interact with objects in the environment by including visual screens and sounds (Bani Mohammadi and Ahmad, 2019). Virtual reality can be defined as a digital simulation created by a computer that allows users to explore a virtual environment and interact with a virtual environment, providing a sense of reality with three-dimensional (3D) images (Bevilacqua et al., 2019). The computer-generated environment helps users experience sensory information such as visual, auditory and movement with experiences close to reality. An important feature of all virtual reality applications is interaction. Virtual environments are created and allow the user to interact not only with the virtual environment, but also with virtual objects in the environment (Bevilacqua et al., 2019; Chirico et al., 2016). Virtual reality, which places people in a central role by using motor skills, decision-making skills, and communication skills with virtual procedures in various clinical environments, is also used as a teaching strategy today (Berman, Durning, Fischer, Huwendiek, & Triola, 2016; Padilha, Machado, Ribeiro, Ramos, & Costa, 2019). Virtual reality simulators are preferred because they increase knowledge retention, clinical reasoning, increased learning satisfaction, and improved motor control, decision-making, and communication skills of individuals and increased self-efficacy (Nassar, Al-Manaseer, Knowlton, & Tuma, 2021; Padilha et al., 2019). Innovations in simulation technologies necessitate the integration of technological developments into health education (Berman et al., 2016). In parallel, the use of high-quality simulators in education strengthens the acquisition of knowledge and skills in students' practices and increases the quality of education (Berman et al., 2016; Padilha et al., 2019).

ELIGIBILITY:
Inclusion Criteria:

* Registered in the midwifery department,
* Attending the normal birth and postpartum period course,
* Agreeing to participate in the study

Exclusion Criteria:

* Having previously taken the normal birth and postpartum period course and failed the course,
* Not attending the episiotomy laboratory course,
* Not agreeing to participate in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2024-12-20 (Actual); Primary Completion 2025-01-10 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
State Anxiety Inventory (STAI) | 1 hours
  The State Anxiety Inventory consists of 20 items and requires the individual to answer how he or she feels at a certain moment and under certain conditions, taking into account his feelings about the situation he is in. The scale is likert type and is a four-degree scale ranging from "Not at all" to "Totally". The maximum score that can be obtained from the scale is 80, and the minimum score is 20. High scores indicate high anxiety, low scores indicate low anxiety.
Episiotomy Self-Efficacy Scale | 1 hours
  The scale developed by the researchers consists of 17 items. The scale is a 5-point Likert type and consists of 4 sub-dimensions. These sub-dimensions are cognitive (5 items), affective (5 items), motivation (3 items) and psychomotor (4 items). The Cronbach Alpha coefficient of this scale developed by the authors is 0.955.

CONTACTS AND LOCATIONS:
Overall Officials: Yasemin Hamlaci Baskaya, Study Director — Sakarya University
Locations (1):
- Sakarya University, Adapazarı, Sakarya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Padilha JM, Machado PP, Ribeiro A, Ramos J, Costa P. Clinical Virtual Simulation in Nursing Education: Randomized Controlled Trial. J Med Internet Res. 2019 Mar 18;21(3):e11529. doi: 10.2196/11529. PMID 30882355
- [Background] Nassar AK, Al-Manaseer F, Knowlton LM, Tuma F. Virtual reality (VR) as a simulation modality for technical skills acquisition. Ann Med Surg (Lond). 2021 Oct 27;71:102945. doi: 10.1016/j.amsu.2021.102945. eCollection 2021 Nov. PMID 34840738
- [Background] Berman NB, Durning SJ, Fischer MR, Huwendiek S, Triola MM. The Role for Virtual Patients in the Future of Medical Education. Acad Med. 2016 Sep;91(9):1217-22. doi: 10.1097/ACM.0000000000001146. PMID 26959224
- [Background] Chirico A, Lucidi F, De Laurentiis M, Milanese C, Napoli A, Giordano A. Virtual Reality in Health System: Beyond Entertainment. A Mini-Review on the Efficacy of VR During Cancer Treatment. J Cell Physiol. 2016 Feb;231(2):275-87. doi: 10.1002/jcp.25117. PMID 26238976
- [Background] Bevilacqua R, Maranesi E, Riccardi GR, Donna VD, Pelliccioni P, Luzi R, Lattanzio F, Pelliccioni G. Non-Immersive Virtual Reality for Rehabilitation of the Older People: A Systematic Review into Efficacy and Effectiveness. J Clin Med. 2019 Nov 5;8(11):1882. doi: 10.3390/jcm8111882. PMID 31694337
- [Background] Bani Mohammad E, Ahmad M. Virtual reality as a distraction technique for pain and anxiety among patients with breast cancer: A randomized control trial. Palliat Support Care. 2019 Feb;17(1):29-34. doi: 10.1017/S1478951518000639. Epub 2018 Sep 10. PMID 30198451
- [Background] Demir-Kaymak Z, Turan Z, Cit G, Akyaman S. Midwifery students' opinions about episiotomy training and using virtual reality: A qualitative study. Nurse Educ Today. 2024 Jan;132:106013. doi: 10.1016/j.nedt.2023.106013. Epub 2023 Oct 31. PMID 37926004
- [Background] Bick DE, Kettle C, Macdonald S, Thomas PW, Hills RK, Ismail KM. PErineal Assessment and Repair Longitudinal Study (PEARLS): protocol for a matched pair cluster trial. BMC Pregnancy Childbirth. 2010 Feb 25;10:10. doi: 10.1186/1471-2393-10-10. PMID 20184764
- [Background] Silf K, Woodhead N, Kelly J, Fryer A, Kettle C, Ismail KM. Evaluation of accuracy of mediolateral episiotomy incisions using a training model. Midwifery. 2015 Jan;31(1):197-200. doi: 10.1016/j.midw.2014.08.009. Epub 2014 Sep 2. PMID 25261381
- [Background] Guler H, Cetin P, Yurtsal ZB, Cesur B, Bekar M, Ucar T, Evcili F, Cetin A. Effect of episiotomy training with beef tongue and sponge simulators on the self-confidence building of midwifery students. Nurse Educ Pract. 2018 May;30:1-6. doi: 10.1016/j.nepr.2018.02.004. Epub 2018 Feb 9. PMID 29452943